CLINICAL TRIAL: NCT05446701
Title: Assessment of Serum FAM19A5 Level in Egyptian Patients With Neuromyelitis Optica Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Khairy Danial, principal investigator, Assiut University
Other Study IDs: Serum FAM9A5 in NMOSD patients
Record Dates: First submitted 2022-04-09; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Assessment of Serum FAM19A5level in Egyptian Patients With NMOSD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 60 case: Sixty patients diagnosed as NMOSD based on the recently revised 2015 international consensus diagnostic criteria for NMOSD (9) ,attending Neurology clinic, Asyut University hospitals, Asyut university and Kasr Al-Ainy multiple sclerosis/neuroimmunology clinic, Cairo University hospitals, Cairo University, Egypt, through one and half year from study onset
  Interventions: Diagnostic Test: serum level of FAM19A5
- 60 control: Sixty healthy volunteers, without any neurological or systemic medical diseases, age and sex matched , will be enrolled as healthy controls(HCs).
  Interventions: Diagnostic Test: serum level of FAM19A5

INTERVENTIONS:
Diagnostic Test: serum level of FAM19A5 — Detection of serum level of FAM19A5 of patients and controls by using ELISA technique.

SUMMARY:
Neuromyelitis optica spectrum disorders (NMOSD) are severe inflammatory autoimmune conditions of the central nervous system (CNS) . The discovery of NMOSD-specific aquaporin 4 (AQP4) antibody has established that NMOSD is indeed a distinct entity . Approximately 80% of patients with NMOSD test positive for aquaporin-4 (AQP4) immunoglobulin G (IgG) antibodies .AQP4-IgG associated NMOSD appears to target astrocytes, not myelin, leading to elevated markers of astrocyte injury during attacks . Untill now there is limited research about understanding the biomarkers of astrocyte injury and the following reactive gliosis. Family with sequence similarity 19-memberA5 (FAM19A5) protein is postulated to regulate nervous and immune cells of the brain as a brain-specific chemokine, but its precise functional role is not well understood . A recent study suggested that FAM19A5 is secreted by reactive astrocytes following CNS damage and triggers reactive gliosis . In another recent study, serum FAM19A5 was higher in patients with NMOSD-AQP4 than in other CNS demyelinating diseases and healthy controls . So, we need to study the level of this novel biomarker among our Egyptian NMOSD patients and whether it shall be a new biomarker for NMOSD .

Moreover just few studies conducted on cognitive dysfunctions in NMOSD patients and they demonstrate a significant decrease of cognitive abilities and the prevalence of CI in different samples varies between 30 and 70% .So further studies are needed to investigate the cognitive performance in NMOSD patients

DETAILED DESCRIPTION:
Sixty patients diagnosed as NMOSD based on the recently revised 2015 international consensus diagnostic criteria for NMOSD ,attending Neurology clinic, Asyut University hospitals, Asyut university and Kasr Al-Ainy multiple sclerosis/neuroimmunology clinic, Cairo University hospitals, Cairo University, Egypt, through one and half year from study onset. Sixty healthy volunteers, without any neurological or systemic medical diseases, age and sex matched , will be enrolled as healthy controls(HCs).

Aim of the work :

1. Determining the serum level of FAM19A5 in a cohort of Egyptian patients with NMOSD in comparison with healthy controls and its relationship with the different clinical phenotypes and parameters and disease severity of NMOSD patients.
2. Cognitive performance of NMOSD patients in comparison with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* 1-Both NMOSD AQP-4 +ve and AQP-4 -ve. 2-Age <18 and >60 years. 3-Both males and females. 4-Both receiving or not receiving current immunosuppressants. 5-Any score of extended disability status scale (EDSS).

Exclusion Criteria:

* 1-Any neuropsychiatric disorder other than NMOSD such as multiple sclerosis ,CNS infectious diseases or malignancy.

  2-Systemic conditions influencing analysis of clinical and serological data , such as general infection, malignancy, and hematologic diseases.

  3-Illiterate patients. 4-History of drug or alcohol abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sixty patients diagnosed as NMOSD based on the recently revised 2015 international consensus diagnostic criteria for NMOSD ,attending Neurology clinic, Asyut University hospitals, Asyut university and Kasr Al-Ainy multiple sclerosis/neuroimmunology clinic, Cairo University hospitals, Cairo University, Egypt, through one and half year from study onset. Sixty healthy volunteers, without any neurological or systemic medical diseases, age and sex matched , will be enrolled as healthy controls(HCs).
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Determining the serum level of FAM19A5 in NMOSD bpatients in relation to healthy controls by using ELISA technique | one and half year
  Determining the serum level of FAM19A5 in NMOSD patients in relation to healthy controls by using ELISA technique

SECONDARY OUTCOMES:
Episodic verbal learning and memory of patients and controls will be evaluated by using California verbal learning test second edition | one and half year
  California verbal learning test second edition (CVL ll)of patients and controls The median of each scale will be assessed for patients and age and sex matched healthy controls on the other side and the impairment will be assessed by comparison

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy EL tellawy, doctorate, Principal Investigator — Assiut University; Nein Shalaby, doctorate, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meng H, Xu J, Pan C, Cheng J, Hu Y, Hong Y, Shen Y, Dai H. Cognitive dysfunction in adult patients with neuromyelitis optica: a systematic review and meta-analysis. J Neurol. 2017 Aug;264(8):1549-1558. doi: 10.1007/s00415-016-8345-3. Epub 2016 Dec 1. PMID 27909800
- [Background] Lee HL, Seok HY, Ryu HW, Cho EB, Kim BC, Kim BJ, Min JH, Seok JM, Shin HY, Kang SY, Kwon OH, Lee SS, Oh J, Sohn EH, Huh SY, Cho JY, Seong JY, Kim BJ. Serum FAM19A5 in neuromyelitis optica spectrum disorders: Can it be a new biomarker representing clinical status? Mult Scler. 2020 Nov;26(13):1700-1707. doi: 10.1177/1352458519885489. Epub 2019 Nov 4. PMID 31680620